CLINICAL TRIAL: NCT01196143
Title: Non-interventional Observational Study to Evaluate the Baseline FSH, Ovarian Volume and AFC (Antral Follicle Count) as Prognostic Factors of the Outcome of the In-vitro Fertilization/Intracytosolic Sperm Injection (IVF/ICSI) in Infertile Patients Who Receive r-FSH (GONAL-f®) for Controlled Ovarian Hyperstimulation
Brief Title: A Study to Evaluate the Baseline Follicle Stimulating Hormone, Ovarian Volume and Antral Follicle Count as Prognostic Factors of the Outcome of In-vitro Fertilisation/Intracytosolic Sperm Injection in Infertile Patients Receiving Gonal f for Controlled Ovarian Hyperstimulation
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 700623-503
Record Dates: First submitted 2010-04-19; First posted 2010-09-08 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: Ovulation induction; Intrauterine insemination; Gonal-f; Controlled ovarian stimulation; Female infertility
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine

SUMMARY:
This is a phase IV non-interventional, multicentric observational study to evaluate the baseline follicle stimulating hormone (FSH) levels, ovarian volume, antral follicle count (AFC) and age as prognostic factors of the outcome of the in-vitro fertilisation/intracytosolic sperm injection (IVF/ICSI) in infertile subjects receiving Gonal-f for controlled ovarian hyperstimulation (COH).

DETAILED DESCRIPTION:
Treatment of subfertility and infertility by assisted reproduction technologies (ART) such as IVF and embryo transfer (ET) requires multiple follicular development to increase the number of female gametes, and the chances of a successful treatment outcome. These technologies include the stimulation of multiple follicular development by exogenous FSH administration and the suppression of endogenous luteinizing hormone (LH) secretion by administration of a GnRH analogue (antagonist or agonist, as required). A single dose of human chorionic gonadotropin (hCG) is administered to mimic the endogenous LH surge and induce final oocyte maturation after adequate follicular development. Recombinant-hFSH (r-hFSH) has been shown to be efficacious in terms of number of oocytes recovered and in terms of pregnancy rates as compared to urinary-hFSH.

Gonal-f fill-by-mass is available as a liquid formulation that can be administered with the pen device. The pen device is prefilled and hence the subject does not require to assemble the device making it simpler to use. The prefilled pen allows the accurate delivery of a precise dose of r-hFSH in 37.5 International Units (IU) increments.

OBJECTIVES

Primary objective:

* Evaluation of the significance of baseline FSH, ovarian volume and AFC with a model adjusted for age as prognostic factors of the IVF/ICSI treatment outcome.

This study planned to enrol 500 female subjects undergoing COH for IVF/ICSI-treatment with Gonal-f. Gonal-f will be administered daily subcutaneously (s.c.) according to the centre's usual clinical practice, commencing on Days 2 or 3 of the cycle during the stimulation period. Treatment with Gonal-f will be continued until adequate follicular development has been achieved with the dose adjusted according to the subject's response, to usually not higher than 450 IU daily. A single injection of 250 micrograms r-hCG or 5,000 IU up to 10,000 IU hCG would be administered 24-48 hours after the last Gonal-f injection to induce final follicular maturation. Gonal-f will be started approximately 2 weeks after the start of an gonadotrophin-releasing hormone (GnRH) agonist treatment, both being continued until adequate follicular development will be achieved. Oocyte retrieval will be done 34-36 hours after hCG administration followed by IVF/ICSI treatment according to clinic's protocol. Each enrolled subject would be followed up until the confirmation of her pregnancy status. Active follow up of all pregnancies will be performed, including those subjects withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female subjects aged between 20-43 years
* Subjects requiring treatment with recombinant FSH for COH for IVF and/or ICSI
* Subjects who are able to communicate well with the investigator and can comply with the requirements of the entire study
* Subjects who have given written informed consent, prior to treatment, with the understanding that consent may be withdrawn by the subject at any time without prejudice

Exclusion Criteria:

* Female subjects not pregnant or lactating
* Subjects with known allergic reaction against one of the ingredients
* Subjects with enlarged ovaries or cysts unrelated to polycystic ovarian disease.
* Subjects with gynaecological bleeding of unknown origin
* Subjects with ovarian, uterine, or mammary cancer
* Subjects with hyperprolactinaemia
* Subjects with tumors of the hypothalamus or the pituitary gland

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects undergoing COH for IVF/ICSI-treatment with Gonal-f in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Up to 28 days after birth

SECONDARY OUTCOMES:
Pregnancy rate (ongoing, clinical, biochemical) | up to 40 weeks post embryo-transfer
  Biochemical: up to 2 weeks post embryo-transfer / clinical: up to 12 weeks post embryo-transfer / ongoing: up to 40 weeks post embryo-transfer
Fertilization rate | 24 hours post oocyte retrieval
Implantation rate | 2 weeks post embryo-transfer
Detailed record of adverse events | Up to 1 year after subject enrollment
Hormone (E2) levels on hCG day | Up to 12 hours prior to hCG administration
Duration of treatment | Up to 12 hours post last FSH injection
Total amount of FSH administered | Up to 1 hour post last FSH injection
Number of oocytes | Up to 1 hour post oocyte retrieval
Miscarriage rate | Up to 12 weeks post embryo-transfer

CONTACTS AND LOCATIONS:
Overall Officials: Michalis Arvanitis, MD, MSc, Study Director — Merck A.E. Hellas,Greece, an affiliate of MerckKGaA, Darmstadt, Germany
Locations (1):
- Centre of Assisted Reproduction "Embryoland", Athens, Greece